CLINICAL TRIAL: NCT06627140
Title: Influence of Expected and Actual Preterm-Birth and Parental Distress on Children's Mental Health 6-11 Years Postpartum
Brief Title: Expected and Actual Preterm-Birth and Parental Distress: Impact on Children's Mental Health
Status: Recruiting | Type: Observational
Sponsor: Goethe University (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Katharina Szota, Dr., Principal Investigator, Goethe University
Other Study IDs: Preterm-Birth & Mental Health
Record Dates: First submitted 2024-09-27; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Preterm Birth; Psychological Distress; Mental Health; Cognitive Functioning
MeSH Terms: conditions — Premature Birth; Psychological Well-Being | interventions — Diagnostic Techniques and Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Risk group: Risk for preterm birth, but no actual preterm birth
  Interventions: Diagnostic Test: Diagnostic procedures
- Preterm birth group: Risk for preterm birth and actual preterm birth
  Interventions: Diagnostic Test: Diagnostic procedures
- Control group: Term birth without risk for preterm birth
  Interventions: Diagnostic Test: Diagnostic procedures

INTERVENTIONS:
Diagnostic Test: Diagnostic procedures — Self- and parent-report on behavioral/emotional symptoms and assessment of cognitive functioning

SUMMARY:
The purpose of the present study is the assessment of the mental health and cognitive development of children 6-11 years after premature or term birth. Impairments in children's' mental health are assessed focusing different disorders or problems (ADHD, Autism traits, Affective disorders, oppositional-aggressive behavior) and using both questionnaires and a clinical interview. Risk and protective factors will be analyzed, e.g., threat and/or actual premature birth compared to term birth, parents' mental health, positive coping, personality traits and social support in the peripartum period and afterwards, as well as medical parameters. The potential interaction of premature birth, medical complications, parental distress and children's mental health will be taken into consideration.

DETAILED DESCRIPTION:
A follow-up survey is conducted based on a previous study on psychological distress in parents with preterm infants (NCT01974531). Medical records and previous questionnaire data will be used for grouping the children based on threat of preterm birth, actual preterm birth and term birth as well as to assess the risk and protective factors in the peripartum period.

Parents have been informed within the first study part that a second study part, including their children, would have been followed. Parents were recontacted and asked for participation via telephone or email. Those who agreed, will be contacted via questionnaires in a first step and then in a second step interviewed regarding their own and their children's mental health. The investigators use the following questionnaires to assess children's mental health: Child Behaviour Checklist 6-18R (CBCL 6-18R), Conners 3rd Edition, Social Communication Questionnaire (SCQ), Revised Children's Anxiety and Depression Scale (RCADS). In addition, the investigators conduct clinical interviews with parents on their children's mental health and assess children's cognitive competencies using the Wechsler Intelligence Scale for Children (WISC-V). The following questionnaires are used to assess parental risk and protective factors: State-Trait Anxiety-Depression Inventory (STADI), Parental Stress Scale (PSS), Parenting Scale Short Form (PS), Big Five Inventory Short Form (BFI).

ELIGIBILITY:
Children and their parents must have participated in the previous study. Inclusion criteria of the previous study regarding the parents were:

* Pregnant women and their partners from the 24th week of gestation on
* 18 years of age

Exclusion criteria of the previous study were:

* Psychiatric, mainly psychotic diseases
* Drug abuse
* Severe neurological disorders
* Stillbirth

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and their parents will be included that participated in the previous study (see above). The study included pregnant women either with risk of preterm birth and term or actual preterm birth from the obstetric ward or a control group without risk from the antenatal class of the obstetric department and their partners.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Children's mental health | Single assessment in Summer/Autumn 2024
  Child Behaviour Checklist 6-18R (CBCL 6-18R), eight problem scales: anxious/depressed (scores from 0 to 26), depressed (scores from 0 to 16), somatic complaints (scores from 0 to 22), social problems (scores from 0 to 22), thought problems (scores from 0 to 30), attention problems (scores from 0 to 20), rule-breaking behaviour (scores from 0 to 34), aggressive behaviour (scores from 0 to 36) with higher scores indicating more difficulties.

SECONDARY OUTCOMES:
Children's cognitive competencies | Single assessment in Autumn/Winter 2024
  Wechsler Intelligence Scale for Children (WISC-V): Composite score on a IQ standard scores. Higher scores indicate a higher overall intellectual ability.

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Szota, PhD, Principal Investigator — Johann Wolfgang Goethe University, Philipps-University Marburg; Susan Schwarz, PhD, Principal Investigator — Goethe University; Silvia Oddo-Sommerfeld, PhD, Principal Investigator — Johann Wolfgang Goethe University Hospital; Frank Louwen, Prof, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Johann Wolfgang Goethe University, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No